CLINICAL TRIAL: NCT06794931
Title: Randomized Pilot Study on the Impact of a Modified Mediterranean Diet (DMM) on the Intestinal Microbiota and Clinical Outcome in Patients With Colorectal Cancer Undergoing Active Medical Oncology Treatment
Brief Title: Study on the Impact of a Modified Mediterranean Diet, in Patients With Colorectal Cancer Undergoing Active Medical Oncology Treatment
Acronym: MIC-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria della Brianza (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MIC-1
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Undefined
Keywords: Colorectal Cancer Metastatic; modified Mediterranean diet; Intestinal microbiota
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified Mediterranean diet (DMM) (Experimental): It consists of a food plan in favor of bacterial biodiversity which focuses above all on foods containing high quality prebiotic fibres, instead reducing the total quantity of fibers compared to the indications provided by the Reference Intake Levels of Nutrients and Energy (LARN) for the Italian population, in consideration of the gastrointestinal side effects of chemotherapy.
  Interventions: Other: Nutrition; Other: Biological samples collection
- standard western diet (DSO) (Other): The Western Diet or standard diet represents the diet most commonly used by the population in many developed countries; it reflects participants' daily eating habits, ensuring that the control group accurately represents typical eating behavior.
  Interventions: Other: Biological samples collection

INTERVENTIONS:
Other: Nutrition — The patient will be instructed to follow the modified Mediterranean diet or his usual diet based on the assigned treatment group.
  Other Names: Specific diet
  Arms: modified Mediterranean diet (DMM)
Other: Biological samples collection — Additional biological samples will also be collected.
  Other Names: Microbiota analyses

SUMMARY:
The study plans to evaluate the impact of the Modified Mediterranean Diet on the biodiversity of the intestinal microbiota (the set of physiological bacteria present at the intestinal level) in patients suffering from metastatic colorectal cancer undergoing chemotherapy treatment +/- biological agent, comparing the microbiota with that of patients following a Western or standard diet.

Specifically, as well demonstrated in clinical studies, there are populations of bacteria that play a role in protecting the intestinal barrier and whose proliferation could be promoted by the Modified Mediterranean Diet.

The study also intends to evaluate the influence of the microbiome on the clinical progress of the disease in terms of side effects and quality of life.

DETAILED DESCRIPTION:
The study will be divided into:

* Screening visit (V0) and Baseline visit (V1): during a control visit, the patient will be asked to participate in the study. After signing the written informed consent for participation in the MIC-1 study, the patient will be screened for his nutritional status. During the visit, a folder will be used to assess nutritional status. Routine blood tests will be carried out, a serum sample will be taken to measure nutritional markers and lifestyle will be assessed. Furthermore, the detection of anthropometric measurements (weight, height, BMI), bioimpedance analysis, estimation of calorie-protein needs and Malnutrition Universal Screening Tool (MUST) nutritional screening is envisaged. Once the study inclusion criteria are met, the patient will return for a visit and randomization into the study arms will take place. Arm A will then be given the modified Mediterranean diet (DMM), while arm B will continue to follow its usual diet. The patient will deliver the fecal sample. Subsequent patient visits will take place every 15 or 21 days depending on the ongoing therapy.
* Visit V2: this visit will be carried out approximately 45 days after the baseline visit. The patient will deliver the stool sample.
* Visit V3: this visit will be carried out approximately 90 days after the baseline visit. During this visit, as per clinical practice, the radiological re-evaluation will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status (ECOG): 0 or 1;
* Age ≥ 18;
* Diagnosis of metastatic colorectal cancer, documented histologically and radiologically according to RECIST 1:1 criteria;
* 1st line chemotherapy treatment +/- biological agent (anti-EGFR, anti-VEGF);
* MUST score 0/1;
* Written informed consent.

Exclusion Criteria:

* Previous oncological medical therapies;
* Indication for parenteral and/or enteral nutrition;
* MUST score > 2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2028-07-23 (Estimated); Study Completion 2028-07-23 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of the modified Mediterranean diet (DMM, Arm A) compared to a standard Western diet (DSO, Arm B) on microbiota | V2 (45 days after V1)
  Comparison of the Firmicutes/Bacteroidetes ratio after 45 days (V2) of first-line chemotherapy +/- biological agent (anti-Epidermal Growth Factor Receptor (EGFR), anti-VEGF) in patients on a modified Mediterranean diet (DMM) compared to patients on a standard Western diet (DSO)

SECONDARY OUTCOMES:
Comparison of the percentage of patients with gastrointestinal effects | V2 (45 days after V1)
  Comparison of the percentage of patients with gastrointestinal effects in Arm A versus Arm B.
Comparison of the percentage of patients with severe gastrointestinal effects | V2 (45 days after V1)
  Comparison of the percentage of patients with severe gastrointestinal effects (G3/G4) in Arm A versus Arm B.
Variation of the change in the Firmicutes/Bacteroidetes ratio | Baseline (V1), after 45 day from baseline (V2), after 90 days from baseline (V3)
  Evaluation of the change in the Firmicutes/Bacteroidetes ratio over 3 time points
Variation of the overall composition of the microbiome | Baseline (V1), after 45 day from baseline (V2), after 90 days from baseline (V3)
  Evaluation of the overall composition of the microbiome over 3 time points
Variation of the microbiome and metabolome | Baseline (V1), after 45 day from baseline (V2), after 90 days from baseline (V3)
  Evaluation of the microbiome and metabolome over 3 time points

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. di Oncologia di Vimercate, ASST-Brianza, Vimercate, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Artale S, Filiali F, Beretta E, Arosio F, Cazzaniga F, Tersalvi C, Sofia M, Tagliabue P, Pozzi P, Colombo A, Carbone C, Pietrogiovanna L, Verga M, Nova P, Calori R, Renso R, Rota S, Aglione S, Manfrida I, Facendola G, Trojani A, Dazzani MC, Basciani S, Valsecchi MG, Capitoli G, Cocola C, Consolandi C. The Effects of a Modified Mediterranean Diet on Gut Microbiota and Chemotherapy Side Effects in Patients With Metastatic Colorectal Cancer Undergoing First-Line Chemotherapy With or Without Either Antiepidermal Growth Factor Receptor or Antivascular Endothelial Growth Factor Agent: Protocol for a Randomized Pilot Study in Italy. JMIR Res Protoc. 2025 Nov 14;14:e72950. doi: 10.2196/72950. PMID 41236788